CLINICAL TRIAL: NCT02913131
Title: Hyperpolarized C-13 Pyruvate as a Biomarker of PI3K/mTOR Pathway Inhibition in Patients With Advanced Solid Tumor Malignancies
Brief Title: Hyperpolarized C-13 Pyruvate as a Biomarker in Patients With Advanced Solid Tumor Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: Rahul Aggarwal (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Rahul Aggarwal, Assistant Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 159517; R01CA183071 (NIH); NCI-2017-02190 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2016-09-20; First posted 2016-09-23 (Estimated); Results first posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pyruvic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Feasibility Run-In (Experimental): Patients with advanced solid tumor malignancies with at least one liver metastasis will be enrolled with iterative adjustment of coil design to optimize imaging parameters including spatial resolution and signal-to-noise ratio (SNR) of hyperpolarized pyruvate / lactate within the target metastatic lesion(s).
  Interventions: Drug: Pyruvate (13C); Device: MRI
- Part B: Biomarker Cohort (Experimental): Patients with advanced solid tumor malignancies and the presence of at least one liver metastasis amenable to hyperpolarized C-13 pyruvate metabolic MR imaging who are planning on being treated with agent targeting PI3K/mTOR pathway will be enrolled.
  Interventions: Drug: Pyruvate (13C); Device: MRI

INTERVENTIONS:
Drug: Pyruvate (13C) — Pyruvate injection followed by an MRI scan.
Device: MRI — MRI scan following the pyruvate (13c) injection

SUMMARY:
This is a single center prospective imaging study investigating the utility of hyperpolarized C-13 pyruvate as a Biomarker of PI3K/mTOR pathway inhibition in patients with advanced solid tumor malignancies. The current protocol will serve as a companion imaging biomarker study paired with therapeutic trials of PI3K/mTOR pathway inhibitors (e.g. CUDC-907, BYL719), as well as a stand-alone protocol for patients treated with standard-of-care therapies inhibiting the PI3K/mTOR signaling pathway (eg. everolimus).

DETAILED DESCRIPTION:
This is a single center prospective imaging study investigating the utility of hyperpolarized C-13 pyruvate/metabolic magnetic resonance (MR) imaging. The current protocol will serve as a companion imaging biomarker study paired with therapeutic trials of PI3K/mTOR pathway inhibitors (e.g. CUDC-907, BYL719), as well as a stand-alone protocol for patients treated with standard-of-care therapies inhibiting the PI3K/mTOR signaling pathway (eg. everolimus).

In Part A (run-in feasibility phase), patients will undergo imaging at a single time point, without paired tumor biopsy. There will be no follow up imaging or requirement for treatment with PI3K/mTOR pathway inhibitor. Iterative adjustment of radiofrequency coil geometry and imaging sequences will be undertaken to optimize intra-tumoral hyperpolarized pyruvate/lactate signal-to-noise ratio.

In Part B, patients will undergo paired baseline hyperpolarized C-13 pyruvate imaging + tumor biopsy,then initiate treatment with agent inhibiting the PI3K/mTOR pathway. After 21 days (+/- 14 days), patients will undergo repeat hyperpolarized C-13 pyruvate MR imaging + tumor biopsy. Patients will subsequently be treated with PI3K/mTOR pathway inhibitor until disease progression, unacceptable toxicity, or patient/physician decision to discontinue therapy.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one target liver or other intra-abdominal lesion detected by standard staging scans that, in the judgment of Study Investigators, would be amenable to hyperpolarized C-13 pyruvate/metabolic MR imaging: Target lesion must measure >=1.0 cm in long axis diameter on CT or MRI
* The subject is able and willing to comply with study procedures and provide signed and dated informed consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Adequate organ function, including creatinine < 1.5 x ULN or estimated creatinine clearance >=500 mL/min (by the Cockcroft Gault equation) and total bilirubin <3x upper limit of normal (ULN).

Part B only:

* No prior local therapy to target lesion.
* If patient agrees to optional biopsy:

  * Presence of at least one target lesion amenable to percutaneous tumor biopsy in the judgment of Interventional Radiology
  * No history of bleeding diathesis.
  * Patients on anti-coagulation they must be able to safely stop treatment for purposes of tumor biopsy.
* Planned treatment with agent targeting PI3K/mTOR pathway (either standard of care or investigational agent)

Exclusion Criteria:

* Patients who because of age, general medical or psychiatric condition, or physiologic status cannot give valid informed consent.
* Patients unwilling or unable to undergo MR imaging, including patients with contra-indications to MRI, such as cardiac pacemakers or non-compatible intracranial vascular clips.
* Metallic implant or device that distorts local magnetic field and compromises the quality of MR imaging.
* Poorly controlled hypertension, defined as systolic blood pressure at study entry greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg. The addition of anti-hypertensives to control blood pressure is allowed.
* Congestive heart failure or New York Heart Association (NYHA) status ≥ 2.
* A history of clinically significant EKG abnormalities, including QT prolongation (QTcF > 500 ms), a family history of prolonged QT interval syndrome, or myocardial infarction (MI) within 6 months of study entry. Patients with rate-controlled atrial fibrillation/flutter will be allowed on study.
* Any condition that, in the opinion of the Principal Investigator, would impair the patient's ability to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in the feasibility cohort (Part A) who completed the scan were permitted the option to enroll in the Biomarker cohort (Part B).
Groups:
- Part B: Biomarker Cohort: Patients with advanced solid tumor malignancies and the presence of at least one liver metastasis amenable to hyperpolarized C-13 pyruvate metabolic magnetic resonance (MR) imaging who are planning on being treated with agent targeting phosphatidylinositol 3-kinase (PI3K)/Mechanistic target of rapamycin (mTOR) pathway will be enrolled.
Period: Overall Study
Arm/Group | Part A: Feasibility Run-In | Part B: Biomarker Cohort
Started | 18 | 5 (Two of the five participants enrolled in Part B were previously enrolled in Part A.)
Completed | 18 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Two of the five participants enrolled in Part B were previously enrolled in Part A.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Feasibility Run-In | Part B: Biomarker Cohort | Total
Number analyzed (Participants) | 18 | 5 | 23
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 1 | 0 | 1
  40-49 years old | 2 | 0 | 2
  50-59 years old | 5 | 1 | 6
  60-69 years old | 4 | 1 | 5
  70-79 years old | 6 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 2 | 15
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 5 | 22
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 2 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 5 | 23

OUTCOME MEASURES:

1. Primary Outcome: Signal-to-noise Ratio (Part A)
Description: The Signal-to-noise ratio with respect to intra-tumoral hyperpolarized (HP) C-13 Lactate/Pyruvate (lac/pyr) ratio detected within target liver or other intra-abdominal metastasis in patients with advanced solid tumor malignancies enrolled in the feasibility cohort will be determined
Time Frame: 1 day
Population: Data for this endpoint was not collected
Arm/Group | Part A: Feasibility Run-In
Number analyzed (Participants) | 0

2. Primary Outcome: Mean Percent Change From Baseline in Peak Intra-tumoral Hyperpolarized Lactate/Pyruvate Ratio (Part B)
Description: Descriptive statistics will be used to characterize the mean change from baseline in intra-tumoral HP pyruvate/lactate ratio after initiation of treatment with PI3K/mTOR pathway inhibitor for participants enrolled in the biomarker cohort, along with 95% confidence interval.
Time Frame: Up to 24 months
Population: Data was not collected for this endpoint for participants in Cohort B
Arm/Group | Part B: Biomarker Cohort
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Reported Treatment-related Adverse Events
Description: Number of participants with documented treatment-related adverse events will be reported for all patients having received a single dose of HP C-13 pyruvate. The study will use the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4 for reporting of adverse events that occur within 3 days of each imaging procedure over the course of the study and any biopsy-related adverse events.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Feasibility Run-In | Part B: Biomarker Cohort
Number analyzed (Participants) | 18 | 5
Participants | 0 | 0

4. Secondary Outcome: Association Between Percent Change From Baseline in Peak Intra-tumoral Hyperpolarized Lactate/Pyruvate Ratio on Metabolic MR Imaging With Clinical Benefit Rate (Part B)
Description: For the purposes of analyzing the association between percent change from baseline in intra-tumoral peak lactate/pyruvate ratio on HP MRI with subsequent clinical outcomes, the cohort will be dichotomized by the median percent change. The objective response rate by RECIST 1.1 criteria and clinical benefit rate (response or stable disease for > 24 weeks) will be compared between dichotomized groups using the chi-squared test.
Time Frame: Up to 24 months
Population: Data was not collected for this endpoint
Arm/Group | Part B: Biomarker Cohort
Number analyzed (Participants) | 0

5. Secondary Outcome: Association Between Percent Change From Baseline in Peak Intra-humoral HP Lactate/Pyruvate Ratio on Metabolic MR Imaging With Progression-free Survival (Part B)
Description: The cohort will be dichotomized by the median percent change. The log-rank test statistic will then be used to test the association of estimates of the hazard functions of the two groups at each observed event time by computing the observed and expected number of events in one of the groups at each observed event time and then adding these to obtain an overall summary across all-time points where there is an event.
Time Frame: Up to 24 months
Population: Data was not collected for this endpoint
Arm/Group | Part B: Biomarker Cohort
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 24 months
Arm/Group | Part A: Feasibility Run-In | Part B: Biomarker Cohort
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/5
Other Adverse Events (participants affected / at risk) | 0/18 | 0/5

LIMITATIONS AND CAVEATS:
The study was closed earlier than expected due to low enrollment in both cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT02913131/Prot_SAP_001.pdf
  • Informed Consent Form (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT02913131/ICF_000.pdf